CLINICAL TRIAL: NCT03152331
Title: Nurse and Physician Stress Reduction: Learning Receptive Awareness Via EEG Feedback
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: C. Michael Dunham (Other)
Collaborators: St. Elizabeth Youngstown Hospital (Unknown)
Responsible Party: Sponsor-Investigator, C. Michael Dunham, Research Associate, Mercy Health Ohio
Organization: Mercy Health Ohio (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-006
Record Dates: First submitted 2017-05-01; First posted 2017-05-15 (Actual); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Stress; Stress, Psychological; Electroencephalography
Keywords: Neurofeedback
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Intervention Model Description: All participants will receive receptive awareness training with neurofeedback.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Receptive Awareness Training (Experimental)
  Interventions: Behavioral: Receptive Awareness Training

INTERVENTIONS:
Behavioral: Receptive Awareness Training — Two 12-minute learning sessions will be conducted for each learning day. Separate instructions will be provided before session 1 and before session 2 to facilitate receptive awareness. The participant is seated in front of a BIS monitor and learns that the BIS number will decrease when in a state of receptive awareness. The trainee will learn to use attentional flexibility in daily activities and adopt willful attention (focal concentration) alternatively with receptive awareness (relaxed attention), as a situation dictates.

SUMMARY:
The purpose of this study is to evaluate a model of mindfulness and neurofeedback among physicians and nurses. Several hypotheses will be tested: 1) BIS values will decrease as the number of sessions increase, 2) wellbeing scores will increase as the number of learning sessions increase, 3) wellbeing scores will be associated with BIS values, and 4) different attentional states will have more or less influence on reducing the BIS value.

DETAILED DESCRIPTION:
For nurses and physicians, concerns exist relative to emotional exhaustion, burnout, and job dissatisfaction. In a study of medical students (median age 25 years), residents/fellows (median age 31 years), and early career physicians (median age 37 years), adverse manifestation rates were 30-40% for emotional exhaustion, 40-50% for burnout, 40-60% for depression, 7-9% for suicidal ideation, and 50-60% for fatigue. The rate of emotional exhaustion, a risk for burnout, has been found to be substantial in nurses in the U.S.

Mindfulness is an attitudinal expression of receptive awareness, wherein there is a distinction made between an experience occurring in the present moment and associated thoughts and interpretations about the experience. The thinking process itself is observed with all thoughts being treated as equal in value, without attraction or rejection. In two investigations that consisted of physicians and nurses, a high mindfulness score was associated with less stress, greater wellbeing, and a positive emotional tone among subjects. Mindfulness training has been associated with reductions in stress or burnout risk in studies that include nurses and physicians.

Neurofeedback (NFB) is a process in which an individual learns to intentionally alter their brainwave activity. NFB has been demonstrated to be useful for decreasing anxiety and enhancing attention.

As concerns with electroencephalographic (EEG) artifacts and the fact that technologies for providing quantitative EEG analysis are continuously evolving, the investigators selected the Bispectral Index (BIS) monitor (Aspect Medical Systems, Newton, MA) as a device to provide NFB signals. The Food and Drug Administration classifies the BIS monitor as an EEG monitoring device that monitors EEG signals, and it may be used for monitoring the effects of anesthetic and sedating agents. The credibility and validity of the device is supported by more than 2,500 citations in the National Library of Medicine that includes publications in the New England Journal of Medicine and Cochrane Systematic Review.

Reductions in BIS values have also been found for conditions other than pharmacologic sedation and include acupressure, stage I sleep, and relaxation using guided imagery.

Although combining mindfulness and NFB has been advocated, such a model, to the investigators' knowledge, has not been evaluated. Therefore, the purpose of the proposed study is to evaluate a model of mindfulness and NFB among physicians and nurses.

ELIGIBILITY:
Inclusion Criteria:

* Physicians (resident, attending, and assistant) at St. Elizabeth Youngstown Hospital
* Nurses (registered, practitioner, and anesthetist) at St. Elizabeth Youngstown Hospital

Exclusion Criterion:

* Individuals undergoing psychological or psychiatric counseling or those requiring psychoaffective medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Bispectral Index Score (BIS) | Up to 28 weeks
  BIS values from baseline to end of study

SECONDARY OUTCOMES:
Wellbeing surveillance tool | Up to 28 weeks
  Wellbeing from baseline to end of study was assessed using the wellbeing surveillance tool, which included elements from the Depression, Anxiety and Stress Scale, Perceived Stress Scale, Positive and Negative Affect Schedule, Medical Outcomes Study Sleep Scale, and Maslach Burnout Inventory
Likert value of each attentional state | Up to 28 weeks
  By computing a mean Likert value for each of four attentional states (all learning days), the effect of each state on reducing the BIS value was rated: 1. widening the visual field, 2. reducing effort, 3. attention to space, and 4. relaxed alertness

CONTACTS AND LOCATIONS:
Overall Officials: C. Michael Dunham, MD, Principal Investigator — St. Elizabeth Youngstown Hospital
Locations (1):
- St. Elizabeth Youngstown Hospital, Youngstown, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dyrbye LN, West CP, Satele D, Boone S, Tan L, Sloan J, Shanafelt TD. Burnout among U.S. medical students, residents, and early career physicians relative to the general U.S. population. Acad Med. 2014 Mar;89(3):443-51. doi: 10.1097/ACM.0000000000000134. PMID 24448053
- [Background] Vahey DC, Aiken LH, Sloane DM, Clarke SP, Vargas D. Nurse burnout and patient satisfaction. Med Care. 2004 Feb;42(2 Suppl):II57-66. doi: 10.1097/01.mlr.0000109126.50398.5a. PMID 14734943
- [Background] Poghosyan L, Clarke SP, Finlayson M, Aiken LH. Nurse burnout and quality of care: cross-national investigation in six countries. Res Nurs Health. 2010 Aug;33(4):288-98. doi: 10.1002/nur.20383. PMID 20645421
- [Background] Perlman DM, Salomons TV, Davidson RJ, Lutz A. Differential effects on pain intensity and unpleasantness of two meditation practices. Emotion. 2010 Feb;10(1):65-71. doi: 10.1037/a0018440. PMID 20141303
- [Background] Atanes AC, Andreoni S, Hirayama MS, Montero-Marin J, Barros VV, Ronzani TM, Kozasa EH, Soler J, Cebolla A, Garcia-Campayo J, Demarzo MM. Mindfulness, perceived stress, and subjective well-being: a correlational study in primary care health professionals. BMC Complement Altern Med. 2015 Sep 2;15:303. doi: 10.1186/s12906-015-0823-0. PMID 26329810
- [Background] Beach MC, Roter D, Korthuis PT, Epstein RM, Sharp V, Ratanawongsa N, Cohn J, Eggly S, Sankar A, Moore RD, Saha S. A multicenter study of physician mindfulness and health care quality. Ann Fam Med. 2013 Sep-Oct;11(5):421-8. doi: 10.1370/afm.1507. PMID 24019273
- [Background] Goodman MJ, Schorling JB. A mindfulness course decreases burnout and improves well-being among healthcare providers. Int J Psychiatry Med. 2012;43(2):119-28. doi: 10.2190/PM.43.2.b. PMID 22849035
- [Background] Kemper KJ, Khirallah M. Acute Effects of Online Mind-Body Skills Training on Resilience, Mindfulness, and Empathy. J Evid Based Complementary Altern Med. 2015 Oct;20(4):247-53. doi: 10.1177/2156587215575816. Epub 2015 Mar 17. PMID 25783980
- [Background] Marzbani H, Marateb HR, Mansourian M. Neurofeedback: A Comprehensive Review on System Design, Methodology and Clinical Applications. Basic Clin Neurosci. 2016 Apr;7(2):143-58. doi: 10.15412/J.BCN.03070208. PMID 27303609
- [Background] Dias AM, van Deusen A. A new neurofeedback protocol for depression. Span J Psychol. 2011 May;14(1):374-84. doi: 10.5209/rev_sjop.2011.v14.n1.34. PMID 21568194
- [Background] Wang JR, Hsieh S. Neurofeedback training improves attention and working memory performance. Clin Neurophysiol. 2013 Dec;124(12):2406-20. doi: 10.1016/j.clinph.2013.05.020. Epub 2013 Jul 1. PMID 23827814
- [Background] Simkin DR, Thatcher RW, Lubar J. Quantitative EEG and neurofeedback in children and adolescents: anxiety disorders, depressive disorders, comorbid addiction and attention-deficit/hyperactivity disorder, and brain injury. Child Adolesc Psychiatr Clin N Am. 2014 Jul;23(3):427-64. doi: 10.1016/j.chc.2014.03.001. PMID 24975621
- [Background] Avidan MS, Zhang L, Burnside BA, Finkel KJ, Searleman AC, Selvidge JA, Saager L, Turner MS, Rao S, Bottros M, Hantler C, Jacobsohn E, Evers AS. Anesthesia awareness and the bispectral index. N Engl J Med. 2008 Mar 13;358(11):1097-108. doi: 10.1056/NEJMoa0707361. PMID 18337600
- [Background] Punjasawadwong Y, Phongchiewboon A, Bunchungmongkol N. Bispectral index for improving anaesthetic delivery and postoperative recovery. Cochrane Database Syst Rev. 2014 Jun 17;2014(6):CD003843. doi: 10.1002/14651858.CD003843.pub3. PMID 24937564
- [Background] Fassoulaki A, Paraskeva A, Kostopanagiotou G, Tsakalozou E, Markantonis S. Acupressure on the extra 1 acupoint: the effect on bispectral index, serum melatonin, plasma beta-endorphin, and stress. Anesth Analg. 2007 Feb;104(2):312-7. doi: 10.1213/01.ane.0000250911.43942.4e. PMID 17242086
- [Background] Dahaba AA, Xue JX, Xu GX, Liu QH, Metzler H. Bilateral Bispectral Index (BIS)-Vista as a measure of physiologic sleep in sleep-deprived anesthesiologists. Minerva Anestesiol. 2011 Apr;77(4):388-93. Epub 2010 Dec 9. PMID 21483382
- [Background] Hudetz JA, Hudetz AG, Reddy DM. Effect of relaxation on working memory and the Bispectral Index of the EEG. Psychol Rep. 2004 Aug;95(1):53-70. doi: 10.2466/pr0.95.1.53-70. PMID 15460358
- [Background] Brandmeyer T, Delorme A. Meditation and neurofeedback. Front Psychol. 2013 Oct 7;4:688. doi: 10.3389/fpsyg.2013.00688. eCollection 2013. No abstract available. PMID 24109463
- [Derived] Dunham CM, Burger AL, Hileman BM, Chance EA, Hutchinson AE, Kohli CM, DeNiro L, Tall JM, Lisko P. Brainwave Self-Regulation During Bispectral IndexTM Neurofeedback in Trauma Center Nurses and Physicians After Receiving Mindfulness Instructions. Front Psychol. 2019 Sep 26;10:2153. doi: 10.3389/fpsyg.2019.02153. eCollection 2019. PMID 31616348
- [Derived] Dunham CM, Burger AL, Hileman BM, Chance EA. Learning receptive awareness via neurofeedback in stressed healthcare providers: a prospective pilot investigation. BMC Res Notes. 2018 Sep 4;11(1):645. doi: 10.1186/s13104-018-3756-0. PMID 30180909